CLINICAL TRIAL: NCT01084122
Title: Efficacy and Safety of Intravenous Iron Sucrose in Patients With Hip Fracture to Prevent Perioperative Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Anna Domingo Trepat, Hospital Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FEIV-DC-09
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-01

CONDITIONS: Hip Fracture; Surgical Intervention
Keywords: Intravenous iron sucrose; Anemia; Transfusion
MeSH Terms: conditions — Hip Fractures; Anemia | interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Iron sucrose — Iron sucrose FERIV® (20 mg/ml). Dilution: 10 ml in 100 ml SF 0.9%. 25 ml in 15 minutes and the rest in others 15 minutes.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intravenous iron sucrose in patients with hip fracture and surgical intervention to prevent perioperative anemia.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the safety and efficacy of intravenous iron sucrose in patients with hip fracture and surgical intervention to prevent perioperative anemia.

It will also determine whether intravenous iron sucrose administration improve outcomes as Haemoglobin values, transfusional needs, postoperative complications, length of hospital stay and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years old
* With Hip fracture or peritrochanteric fracture.
* Who needs surgical intervention.
* And sign the informed consent form.

Exclusion Criteria:

* Tumor pathological fracture.
* Two or more long bone fractures.
* Seric Ferritin levels > 300 ng/ml.
* Hypersensitivity to Iron sucrose or any component of the formulation.
* Patients with allogeneic transfusion rejection.
* Patients with previous blood transfusion request (Hb< 8g/dl).
* Patients treated with hematopoietic growth factors.
* Patients with Anticoagulant treatment, due to thromboembolic high risk disease.
* Asthma in treatment.
* Cirrhosis, Acute Hepatitis, or increased Aminotransferases (> 3 times the upper limit of normal).
* Advanced Dementia (GDS>5) from the Global Deterioration Scale.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Transfusional needs | 1st, 5th day and 1st and 6 th month after surgical intervention.
  Blood transfusion rate in patients over 65 years undergone hip fracture and surgical intervention.

SECONDARY OUTCOMES:
Units of packed cells | 1st and 5th days, 1st and 6th month after surgical intervention.
  Packed cells average.
Postoperative complications | 1st and 5th day , 1st and 6th month after surgical intervention.
  Infections, adverse reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Cirugía Ortopédica y Traumatología. Hospital Clinic., Barcelona, Barcelona, Spain